CLINICAL TRIAL: NCT07090265
Title: Evaluation of The Periodontal Parameters Following Non-Surgical Periodontal Therapy With and Without Adjunctive Use of Injectable Platelet Rich Fibrin: A Randomized Controlled Clinical Trial
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Gulf Medical University (Other)
Responsible Party: Principal Investigator, Mohamed Atef Abd El Moneium, Assistant Professor of Periodontics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-COD-STD-71-FEB-2024
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Periodontitis (Stage 3)
Keywords: Periodontitis; Injectable Platelet Rich Fibrib; Non-surgical Periodontal Therapy; Adjunctive Therapy
MeSH Terms: conditions — Periodontitis | interventions — proliferation regulatory factors, human urine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-surgical Periodontal Therapy (Active Comparator): Non-surgical Periodontal Therapy using ultrasonic scaling and root debridement using Gracey Curettes
  Interventions: Procedure: non-surgical periodontal therapy
- Non-surgical Periodontal Therapy + Injectable Platelet Rich Fibrin (Experimental): Non-surgical Periodontal Therapy using ultrasonic scaling and root debridement using Gracey Curettes with adjunctive use of Injectable Platelet Rich Fibrin
  Interventions: Procedure: non-surgical periodontal therapy + I-PRF

INTERVENTIONS:
Procedure: non-surgical periodontal therapy — Mechanical Root Instrumentation using Ultrasonic scaling and root debridement using Gracey Curettes
  Arms: Non-surgical Periodontal Therapy
Procedure: non-surgical periodontal therapy + I-PRF — Mechanical Root Instrumentation using Ultrasonic scaling and root debridement using Gracey Curettes following by subgingival application of I-PRF
  Arms: Non-surgical Periodontal Therapy + Injectable Platelet Rich Fibrin

SUMMARY:
This randomized controlled clinical trial aims to evaluate the effectiveness of non-surgical periodontal therapy (NSPT) with and without the adjunctive use of injectable platelet-rich fibrin (I-PRF) in patients with chronic periodontitis. The primary objective is to assess changes in key periodontal parameters including probing depth (PD), clinical attachment level (CAL), bleeding on probing (BOP), and plaque index (PI) over a defined follow-up period. Participants will be randomly assigned to two groups: one receiving standard NSPT alone and the other receiving NSPT combined with subgingival application of I-PRF. The study seeks to determine whether the adjunctive use of I-PRF can enhance periodontal healing and improve clinical outcomes compared to conventional therapy alone.

DETAILED DESCRIPTION:
This randomized controlled clinical trial is designed to assess the clinical efficacy of non-surgical periodontal therapy (NSPT) with and without the adjunctive use of injectable platelet-rich fibrin (I-PRF) in the management of chronic periodontitis. Periodontal disease is a multifactorial inflammatory condition characterized by progressive destruction of the supporting structures of the teeth. NSPT, primarily through scaling and root planing (SRP), remains the gold standard for initial therapy. However, the regeneration of periodontal tissues following NSPT can be limited, especially in moderate to advanced cases.

Injectable PRF (I-PRF) is a second-generation autologous platelet concentrate prepared without anticoagulants, offering a fluid formulation rich in platelets, leukocytes, and growth factors. Its injectable nature allows subgingival delivery, promoting enhanced wound healing and soft tissue regeneration. This study aims to investigate whether adjunctive use of I-PRF following SRP can provide superior clinical outcomes compared to SRP alone.

Participants diagnosed with generalized chronic periodontitis, presenting with probing depths ≥5 mm in at least two quadrants, will be enrolled. Subjects will be randomly allocated into two groups:

Test Group: Undergo NSPT (scaling and root planing) followed by subgingival injection of I-PRF at selected sites.

Control Group: Undergo NSPT alone without any adjunctive treatment.

I-PRF will be prepared via low-speed centrifugation of venous blood immediately prior to application and injected subgingivally at the affected sites immediately after completion of SRP.

Clinical parameters including probing depth (PD), clinical attachment level (CAL), bleeding on probing (BOP), and plaque index (PI) will be recorded at baseline and at 3 months post-treatment. All procedures and assessments will be performed by calibrated, blinded examiners.

The primary outcome measure is the change in clinical attachment level at 3 months. Secondary outcome measures include reductions in PD and BOP, and improvements in PI. The study will help determine whether I-PRF can serve as a minimally invasive, biologically driven adjunct to enhance the outcomes of conventional NSPT.

This investigation is expected to contribute to evidence-based decision-making regarding the adjunctive use of autologous biologics in periodontal therapy.

ELIGIBILITY:
Inclusion Criteria:

Medically free, Non-smokers, Stage III Periodontitis Patients, Probing depth <5mm

Exclusion Criteria:

* Systemic disease, Smoking, Pregnancy, History of Chemotherapy, Radiotherapy

Max Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment Gain | 3 months
  the change in the distance from the Cemento-Enamel Junction to the base of the periodontal pockets

SECONDARY OUTCOMES:
Probing Depth Reduction | 3 months
  The change in the distance from the gingival margin to the base of the periodontal pocket
Bleeding on Probing | 3 months
  the response to the walking of the probe on the lateral wall of the periodontal pocket

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Atef, Ph.D., Study Director — Gulf Medical University
Locations (1):
- Gulf Medical University, Ajman, Ajman Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided